CLINICAL TRIAL: NCT06877481
Title: Turkish Adaptation, Validation, and Reliability Assessment of the Geriatric Pain Measure - Short Form
Brief Title: Turkish Validation of the Geriatric Pain Measure - Short Form
Status: Recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Tuba Tanyel Saraçoğlu, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Other Study IDs: 26.02.2025.73
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Geriatric Assessment; Pain Measurement; Chronic Pain
Keywords: Geriatric Assessment; Pain Measurement; Chronic Pain; Geriatric Pain Measurement Short Form
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Geriatric Patients with Chronic Pain: Geriatric patients (≥65 years) with chronic pain who are examined at the Pain Management Clinic of Başakşehir Çam and Sakura City Hospital. Participants will be assessed under the supervision of pain management and gerontology specialists.
  Interventions: Other: Geriatric Pain Measurement Short Form

INTERVENTIONS:
Other: Geriatric Pain Measurement Short Form — Geriatric Pain Measure - Short Form (GPM-SF) is a validated pain assessment tool designed specifically for older adults. It is a 12-item questionnaire that evaluates pain intensity, interference with daily activities, and emotional impact of chronic pain in geriatric patients. The short form provides a quick and reliable assessment of pain-related disability in older populations.

SUMMARY:
This study aims to adapt, validate, and assess the reliability of the Geriatric Pain Measure - Short Form in Turkish. A total of 150 patients aged 65 years and older will complete the scale under the supervision of pain management and gerontology specialists. Reliability and validity will be evaluated using statistical analyses, including internal consistency, test-retest reliability, and correlation with validated pain and sleep scales. Ethical approval has been obtained, and all participants will provide informed consent.

DETAILED DESCRIPTION:
For the Turkish adaptation, validation, and reliability study of the Geriatric Pain Measure - Short Form, permission was obtained from Dr. Eva Blozik, the original developer of the scale. The adaptation process will follow standard cross-cultural validation guidelines, including forward translation into Turkish by an expert group, back-translation into English by a separate expert group, and comparison of the back-translated version with the original English version for conceptual and linguistic accuracy. A multidisciplinary expert panel, including Turkish language specialists and pain management experts, will review the final Turkish version, making necessary cultural adaptations to ensure semantic equivalence. The study will involve 150 patients aged 65 years and older visiting the Pain Management Clinic, where they will complete the Turkish version of the scale under the supervision of pain management and gerontology specialists. Reliability will be assessed through internal consistency (Cronbach's alpha), test-retest reliability, and item-total correlations, while construct validity will be evaluated using factor analysis. Concurrent validity will be examined by correlating the Turkish version of the scale with other outcome measures. Ethical approval has been obtained from Başakşehir Çam and Sakura City Hospital Ethics Committee, and all participants will provide written informed consent before participation.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric patients with chronic pain
* Patients who agreed to participate in the study

Exclusion Criteria:

* Demantia
* Mental of physical disorders that effect patients answering the scales
* Diagnosis of malignancy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 65 years of age who applied to the pain management outpatient clinic with the complaint of chronic pain and consented to participate the study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Geriatric Pain Measurement Short Form | Day 1
  Geriatric Pain Measure - Short Form (GPM-SF) is a validated pain assessment tool designed specifically for older adults. It is a 12-item questionnaire that evaluates pain intensity, interference with daily activities, and emotional impact of chronic pain in geriatric patients. The short form provides a quick and reliable assessment of pain-related disability in older populations.
Numerik Rating Scale | Day 1
  The Numeric Rating Scale (NRS) is a 0 to 10 scale used to assess pain intensity, where 0 = no pain and 10 = worst possible pain. It is a simple, reliable tool widely used in clinical and research settings.
FRAIL Scale | Day 1
  The FRAIL Scale is a five-item questionnaire used to assess frailty in older adults. It evaluates Fatigue, Resistance (weakness), Ambulation (mobility), Illnesses (comorbidities), and Loss of weight. A higher score indicates a greater degree of frailty, helping identify patients at risk for adverse health outcomes.
Lawton & Brody Instrumental Activities of Daily Living Scale | Day 1
  The Lawton & Brody Instrumental Activities of Daily Living, a scale that assesses an older adult's ability to perform eight complex daily tasks essential for independent living. These tasks include using the telephone, shopping, meal preparation, housekeeping, laundry, transportation, medication management, and handling finances. It helps evaluate functional independence and detect early declines in cognitive or physical abilities
Geriatric Depression Scale-15 | Day 1
  The Geriatric Depression Scale-15 (GDS-15) is a shortened version of the original GDS, consisting of 15 yes/no questions designed to screen for depression in older adults. It is simple, quick, and reliable, making it suitable for use in clinical and research settings, including in patients with mild cognitive impairment. Higher scores indicate more depressive symptoms.
Pittsburgh Sleep Quality Index | Day 1
  The Pittsburgh Sleep Quality Index is a self-reported questionnaire assessing sleep quality over the past month. It includes 18 items evaluating aspects such as sleep duration, latency, disturbances, efficiency, daytime dysfunction, and use of sleep medications. A higher total score indicates poorer sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Başakşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No